CLINICAL TRIAL: NCT05657847
Title: Novel Complex Radiodiagnostics of Peripherial Arthropathies
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Collaborators: National Institute of Rheumatology and Physiotherapy, Hungary (Unknown); Buda Hospital of the Hospitaller Order of Saint John of God (Unknown)
Responsible Party: Sponsor
Other Study IDs: IV/664-3/2022/EKU
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-07

CONDITIONS: Arthritis, Rheumatoid; Arthritis, Psoriatic; Crystal Arthropathies
Keywords: photon-counting detector computer tomography, magnetic resonance imaging, radiography, rheumatoid arthritis, psoriatic arthritis, crystal arthropathies
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Crystal Arthropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Rheumatoid arthritis: Rheumatoid arthritis patients. (American College of Rheumatology (ACR) 1987, ACR/European League Against Rheumatism (EULAR) >18 years Imaging studies: CT and X-ray/MRI/US Physical examination by the rheumatologist and laboratory tests which are conventionally necessary for the diagnosis (including RF, ACPA)
  Interventions: Device: Photon-counting detector-CT
- Psoriatic arthritis: Psoriatic arthritis patients. (CASPAR Criteria) >18 years Imaging studies: CT and X-ray/MRI/US Physical examination by the rheumatologist and laboratory tests which are conventionally necessary for the diagnosis.
  Interventions: Device: Photon-counting detector-CT
- Crystal arthropathies: Crystal arthropathies patients. >18 years Imaging studies: CT and X-ray/MRI/US Physical examination by the rheumatologist and laboratory tests which are conventionally necessary for the diagnosis.
  Interventions: Device: Photon-counting detector-CT

INTERVENTIONS:
Device: Photon-counting detector-CT — CT scan

SUMMARY:
Chronic peripherial arthritides are common diseases with soaring public health consequences. Our goal is to assess the role of photon-counting detector computed tomography in the diagnostics of peripherial arthropathies.

DETAILED DESCRIPTION:
Background:

Chronic peripherial arthritides include immune-mediated (rheumatoid arthritis, psoriatic arthritis) and crystal deposition diseases (gout, pseudogout, hydroxiapatite-deposition disease).

Conventional radiographs are utilized to screen arthritis-associated deformities, bone erosions and joint space narrowing. MRI is able to detect bone marrow edema, synovitis and the swelling of soft tissues. Sonography can also detect synovitis and soft tissue involvement but does not provide information about bone marrow edema and poorly assess erosions. Photon-counting detector computed tomography (PCD-CT) is a novel type of CT device which provides many advantages like improved signal-to-noise ratio, intrinsic spectral information, lower radiation exposure, and better spatial resolution. PCD-CT is a type of X-ray computed tomography in which X-rays are detected using a photon-counting detector. These detectors are able to directly transform X-ray photons into electrical signals. Compared to previous generation scintillation detectors, photon-counting detectors have several advantages: being able to count the charges created by individual x-ray photons and measuring their energy level also providing multi- energy spectral sensitivity. 0.2 mm slice thickness potentiates the detection of bone erosionss. Collagen-rich structures like cartilage, ligaments, and tendons are easier to identify on PCD-CT images. Bone marrow edema can be visualized with virtual non- calcium reconstruction. PCD-CT could both detect and differentiate cristal deposits.

Aims: To assess the possible role of PCD-CT technique in the diagnostics of peripherial arthropathies.To compare the role of PCD-CT in the detection of arthritis-related pathologies with other imaging modalities like MRI and conventional radiography.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis (EULAR/ACR Criteria) / Psoriatic arthritis (CASPAR Criteria)/ Crystal arthropathies
* signed informed consent

Exclusion Criteria:

* age: <18 years, > 100 years
* pregnant
* breastfeeding

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults suffering from peripherial arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Bone erosions | From baseline to at least 2 years
  To assess the detection of arthritis-related bone erosions with different imaging techniques, including PCD-CT.
Bone marrow edema and periarticular soft tissue involvement | From baseline to at least 2 years
  To assess the detection of arthritis-related bone marrow edema and periarticular soft tissue with different imaging techniques, including PCD-CT.
Crystal deposit characterization | From baseline to at least 2 years
  To detect the different crystal deposits with PCD-CT.

SECONDARY OUTCOMES:
To evaluate the performance of PCD-CT in the detection of active arthritis-related imaging findings and structural damages. | From baseline to at least 3 years
  To compare the performance of PCD-CT with different modalities in the diagnostics of peripherial arthropathies.

CONTACTS AND LOCATIONS:
Locations (3):
- Hungary (3):
  - National Institute of Rheumatology and Physiotherapy, Budapest
  - Buda Hospital of the Hospitaller Order of Saint John of God, Budapest
  - Semmelweis University, Budapest

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Duryea J, Dobbins JT 3rd, Lynch JA. Digital tomosynthesis of hand joints for arthritis assessment. Med Phys. 2003 Mar;30(3):325-33. doi: 10.1118/1.1543573. PMID 12674232
- [Background] Stamp LK, Anderson NG, Becce F, Rajeswari M, Polson M, Guyen O, Viry A, Choi C, Kirkbride TE, Raja AY. Clinical Utility of Multi-Energy Spectral Photon-Counting Computed Tomography in Crystal Arthritis. Arthritis Rheumatol. 2019 Jul;71(7):1158-1162. doi: 10.1002/art.40848. Epub 2019 May 28. PMID 30714678
- [Background] Adams JE, Chen SZ, Adams PH, Isherwood I. Measurement of trabecular bone mineral by dual energy computed tomography. J Comput Assist Tomogr. 1982 Jun;6(3):601-7. doi: 10.1097/00004728-198206000-00028. PMID 7096705
- [Background] Woodworth TG, Morgacheva O, Pimienta OL, Troum OM, Ranganath VK, Furst DE. Examining the validity of the rheumatoid arthritis magnetic resonance imaging score according to the OMERACT filter-a systematic literature review. Rheumatology (Oxford). 2017 Jul 1;56(7):1177-1188. doi: 10.1093/rheumatology/kew445. PMID 28398508
- [Background] Ostergaard M, Ejbjerg B, Szkudlarek M. Imaging in early rheumatoid arthritis: roles of magnetic resonance imaging, ultrasonography, conventional radiography and computed tomography. Best Pract Res Clin Rheumatol. 2005 Feb;19(1):91-116. doi: 10.1016/j.berh.2004.08.006. PMID 15588973
- [Background] Fukuda T, Umezawa Y, Asahina A, Nakagawa H, Furuya K, Fukuda K. Dual energy CT iodine map for delineating inflammation of inflammatory arthritis. Eur Radiol. 2017 Dec;27(12):5034-5040. doi: 10.1007/s00330-017-4931-8. Epub 2017 Jul 3. PMID 28674965
- [Background] Mallinson PI, Coupal TM, McLaughlin PD, Nicolaou S, Munk PL, Ouellette HA. Dual-Energy CT for the Musculoskeletal System. Radiology. 2016 Dec;281(3):690-707. doi: 10.1148/radiol.2016151109. PMID 27870622
- [Background] Finkenstaedt T, Manoliou A, Toniolo M, Higashigaito K, Andreisek G, Guggenberger R, Michel B, Alkadhi H. Gouty arthritis: the diagnostic and therapeutic impact of dual-energy CT. Eur Radiol. 2016 Nov;26(11):3989-3999. doi: 10.1007/s00330-016-4237-2. Epub 2016 Feb 4. PMID 26847043
- [Background] Willemink MJ, Persson M, Pourmorteza A, Pelc NJ, Fleischmann D. Photon-counting CT: Technical Principles and Clinical Prospects. Radiology. 2018 Nov;289(2):293-312. doi: 10.1148/radiol.2018172656. Epub 2018 Sep 4. PMID 30179101